CLINICAL TRIAL: NCT00094263
Title: Long-Term Predictors of Morbidity in Older Age
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1273; R21HL075259 (NIH)
Record Dates: First submitted 2004-10-15; First posted 2004-10-15 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Diabetes Mellitus; Heart Diseases; Heart Failure; Heart Failure, Congestive; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Heart Diseases; Heart Failure; Obesity

SUMMARY:
To use existing longitudinal data from the Chicago Heart Association and Western Electric Company studies to examine adiposity in relation to heart failure, multimorbidity and to examine heart rate in relation to incident diabetes.

DETAILED DESCRIPTION:
BACKGROUND:

Obesity is reaching epidemic proportions in the U.S. with over 50 percent of the adult population either overweight or obese. Obesity has been studied extensively as a risk factor for coronary heart disease and stroke, but has received less attention as a risk factor for congestive heart failure (CHF). Another area of limited investigation is the study of risk factors for multi morbidity, i.e. the occurrence of several morbid events at the same time, which is very common in older adults. Other areas of investigation in this study are possible associations between each of heart rate and dietary patterns with the development of diabetes. The Chicago Heart Association Detection Project and the Western Electric studies, both supported by the National Heart, Lung, and Blood Institute, are resources to study the above associations. Multiple measures of obesity are available at several different time points and follow-up data are available for 30-40 years which should increase the power of the study.

Data to be used for this project include baseline data collected in 1967-73 from 39,522 subjects from the Chicago Heart Association Study (CHA) and baseline and annual follow-up data from the Western Electric Study collected from 1957-1966 consisting of 2107 men, age 40-55 years in the Chicago area. Mortality follow-up for those 2 cohorts is accomplished via the National Death Index. Morbidity follow-up is accomplished by record linkage with Medicare files and to some extent by followup questionnaires for disease outcomes although the follow-up rate for the latter approach is only about 60 percent.

DESIGN NARRATIVE:

The study uses extensive existing data from the Chicago Heart Association (CHA) [20,854 men and 16,049 women aged 18-64 at baseline (1967-73)] and Western Electric (WE) [2,107 men aged 40- 55 at baseline (1957-58)] that include four comprehensive sources of outcomes: 1) mortality data from long-term follow-up; 2) morbidity and other data from Medicare claims for 19 years from 1984 to 2000; 3) multiple health questionnaires (CHA); and 4) repeated measures of adiposity from 8 annual re-examinations after baseline (WE). The study addresses the following specific aims: 1) to investigate in-depth the longitudinal associations of adiposity as assessed by several indices (body mass index, weight gain, subscapular and triceps skinfolds, and derived percent body fat) during young adulthood and middle age with mortality and morbidity from congestive heart failure later in life; 2) to delineate the relationships of adiposity assessed earlier in life with older-age multimorbidity, the coexistence of multiple pathological conditions of varying severity -- a very common but under-studied phenomenon among older adults; 3) to examine in-depth the associations of heart rate and changes in heart rate with incident diabetes, stratified by obesity status at baseline. As an exploratory aim, the study will assess whether a) higher fruit and vegetable and lower sugar intake; and b) higher dairy and calcium intake are associated with lower adiposity, smaller weight gain, and lower incidence of diabetes.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lijing Yan — Northwestern University